CLINICAL TRIAL: NCT02276404
Title: Entspannung Und Akupunktur Zur Reduktion Perioperativer Symptome Bei Brustkrebspatientinnen- Eine Randomisiert-kontrollierte Interventionsstudie im Kontext Einer Integrativ Onkologischen Versorgung (EARpeS)
Brief Title: Preoperative Relaxation Training and Acupuncture to Minimize Perioperative Symptoms in Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Silke Lange, Research fellow, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14-5778-BO
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2019-06-14 (Actual); Status verified 2019-06

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Relaxation Therapy; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- relaxation training (Experimental): Each participant of the experimental group 1 receives 2 one-hour sessions of guided relaxation training prior to surgery.
  Interventions: Behavioral: relaxation training
- acupuncture (Experimental): Each participant of the experimental group 2 receives 3 acupuncture treatments with a semi-standardized acupoint scheme: once a week over 2 weeks and the day before surgery.
  Interventions: Other: acupuncture
- relaxation training and acupuncture (Experimental): Each patient of the experimental group 3 receives 3 acupuncture treatments with a semi-standardized acupoint scheme and 2 one-hour sessions of guided relaxation training prior to surgery.
  Interventions: Behavioral: relaxation training; Other: acupuncture
- usual care (No Intervention): Patients receive usual senological treatment

INTERVENTIONS:
Behavioral: relaxation training — The relaxation sessions comprise an introduction in 3 relaxation techniques conducted by a mind-body therapist: "Body Scan", mindfulness meditation and imagination. Patients also receive a CD with different relaxation exercises and the instruction to exercise daily at home for at least 15 minutes.
  Arms: relaxation training; relaxation training and acupuncture
Other: acupuncture — The acupuncture treatment comprises needling of 6 standardized acupoints: Pericardium 6, Stomach 36, Large intestine 4, Spleen/Pancreas 10, Dumai 20, Liver 3, Shenmen. Additional points can be chosen individual.
  Arms: acupuncture; relaxation training and acupuncture

SUMMARY:
Breast cancer surgery is associated with presurgical psychological distress and clinically significant side effects including postsurgical pain, nausea and fatigue. A few studies have examined how to intervene to assist women undergoing breast cancer surgery. For example presurgical hypnosis has been proven to decrease side effects and even intraoperative anesthesia use. Besides the more psychologically based interventions there are a few studies suggesting positive effects of acupuncture on pain, anxiety and nausea in surgery patients.This study aims to investigate whether a presurgical relaxation training, acupuncture treatment or a combination of both therapies is able to reduce presurgical psychological distress an postsurgical side effects in breast cancer patients in comparison to usual care.

ELIGIBILITY:
Inclusion criteria:

* clinically proven breast cancer with an indication for breast conserving surgery with max. 50% volume reduction
* physical and psychological ability to take part in relaxation training

Exclusion criteria:

* serious psychiatric disorder
* to time span to surgery shorter than 2 weeks or longer than 20 weeks

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

PRIMARY OUTCOMES:
presurgical psychological distress | expected average of 13 days
  Measured by 100mm visual analog scale 1 day pre surgery
postsurgical pain | expected average of 15 days
  Measured by 100mm visual analog scale 1 day post surgery

SECONDARY OUTCOMES:
postsurgical psychological distress | expected average of 15 days
  Measured by 100mm visual analog scale 1 day post surgery
postsurgical psychological distress | expected average of 21 days
  Measured by 100mm visual analog scale 1 week post surgery
postsurgical pain | expected average of 21 days
  Measured by 100mm visual analog scale 1 week post surgery
postsurgical nausea | expected average of 15 days
  Measured by 100mm visual analog scale 1 day post surgery
postsurgical nausea | expected average of 21 days
  Measured by 100mm visual analog scale 1 week post surgery
postsurgical fatigue | expected average of 15 days
  Measured by 100mm visual analog scale 1 day post surgery
postsurgical fatigue | expected average of 21 days
  Measured by 100mm visual analog scale 1 week post surgery
intraoperative analgesia use | expected average of 14 days
  intraoperative analgesia use is taken from operative logs
intraoperative anesthesia use | expected average of 14 days
  intraoperative anesthesia use is taken from operative logs
postoperative analgesia use | expected average of 15 days
  postoperative analgesia use is taken from medical records
immunemodulation | expected average of 14 days
  natural killer cell activity is measured at begin of surgery
immunemodulation | expected average of 14 days
  natural killer cell activity is measured at end of surgery
Number of patients with adverse events | expected average of 21 days
  Number of patients with adverse events are measured one week post surgery
presurgical psychological distress | expected average of 13 days
  Measured by Profile of Mood States (POMS) 1 day pre surgery
postsurgical psychological distress | expected average of 15 days
  Measured by Profile of Mood States (POMS) 1 day post surgery
postsurgical psychological distress | expected average of 21 days
  Measured by Profile of Mood States (POMS) 1 week post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gustav J. Dobos, Prof, Study Chair — Chair of Complementary and Integrative Medicine, Universitay of Duisburg-Essen, Germany
Locations (1):
- Department of Senology, Kliniken Essen-Mitte, Essen, Germany